CLINICAL TRIAL: NCT05234489
Title: A Phase 1, Open-label, Dose-ranging Study to Assess the Safety, Tolerability, Preliminary Efficacy, and Dose Effect of Signature Cord Product in Patients With Symptomatic Osteoarthritis of the Knee
Brief Title: Study to Assess Signature Cord Product in Patients With Symptomatic OA of the Knee
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Thomas Klootwyk, MD (Other)
Collaborators: Signature Biologics, LLC (Unknown); KLM Solutions, LLC (Unknown)
Responsible Party: Sponsor-Investigator, Thomas Klootwyk, MD, Orthopedic Surgeon, Forte Sports Medicine and Orthopedics
Organization: Forte Sports Medicine and Orthopedics (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIG001-OAK-01
Record Dates: First submitted 2022-01-07; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis, Knee
Keywords: Allogeneic Umbilical Cord Tissue
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: The Phase 1 trial will enroll 5 subjects into an initial group receiving a low dose of SIG001. Provided that these subjects tolerate this dose well, will proceed to enroll 5 subjects into a group receiving a high dose of SIG001.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low Dosage Group (Active Comparator): This group will receive the lower dose (75mg) of the investigational product.
  Interventions: Biological: Signature Cord Prime
- High Dosage Group (Active Comparator): This group will receive the higher dose (150mg) of the investigational product.
  Interventions: Biological: Signature Cord Prime

INTERVENTIONS:
Biological: Signature Cord Prime — Low dose - Subjects will receive SIG001 (75 mg) which will be diluted to a total of 4 ml volume with Ringer's Lactate.
  High dose - Subjects will receive SIG001 (150mg) which will be diluted to a total of 4 ml volume with Ringer's Lactate.

SUMMARY:
This study is a Phase 1 trial. The overall objective is to evaluate the safety and potential efficacy of a specific type of umbilical cord tissue-derived product (SIG001), which, other than a change in cryopreservation medium to render it compatible with cGMP, is similar to the reported real-world experience from 2 clinics on 135 knees.

DETAILED DESCRIPTION:
Primary Objective:

A Phase 1, open-label, non-controlled trial, to assess the safety of intra-articular injection of SIG001, at either of two doses, in a total of 10 patients with Symptomatic Osteoarthritis of the Knee, Kellgren-Lawrence Grade 2-3, at 7, 30, 90 and 180 days after dosing.

Secondary Objective:

A Phase 1, open-label, non-controlled trial, to obtain very early data relating to any effects of intra-articular injection of SIG001, at either of two doses pain, activity, and quality of life in 10 patients with Symptomatic Osteoarthritis of the Knee, Kellgren-Lawrence Grade 2-3, at 7, 30, 90 and 180 days.

Study Design:

The Phase 1 trial will enroll 5 subjects into an initial group receiving a low dose of SIG001. Provided that these subjects tolerate this dose well, will proceed to enroll 5 subjects into a group receiving a high dose of SIG001.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of osteoarthritis of the knee based on clinical and radiographic findings
* Kellgren-Lawrence Grades 2-3
* Average pain score, on a 100-point numerical rating scale (VAS), over the past 7 days of > 40 and < 90 in the index knee and < 40 in the contralateral knee
* Body mass index < 35 kg/m²
* Ability to comply with the requirements of the study
* Ability to understand and provide written informed consent
* Not suspecting or expecting to be pregnant during the study period
* All participants of reproductive age/capacity to confirm the use of adequate contraception during the study period

Exclusion Criteria:

* Prior therapeutic radiation to the index knee
* Use of any pain medication or therapy less (anticoagulants, non-steroidal anti-inflammatory drugs (NSAIDS) oral and topical, topical CBD, and narcotics) than 15 days prior to test product administration that has not or will not have had a stable dosage, frequency, or intensity for at least 3 months prior to test agent administration. Use of oral NSAIDs at a stable dose at least 3 months prior to test agent administration must be continued through the study period.
* Intra-articular treatment with corticosteroids, regenerative medicines (e.g., plasma, stem cell, placental products), or systemic steroid use within 3 months prior to screening
* Intra-articular treatment with hyaluronic acid within 6 months prior to screening
* Surgical intervention on the index knee < 12 months, or arthroscopy < 3 months prior to screening
* Non-ambulatory status
* Past or current diagnosis of fibromyalgia or inflammatory arthritis, gout, rheumatoid arthritis, lupus arthropathy, psoriatic arthritis, avascular necrosis, severe bone deformity, active infection of the index knee joint or at the site of injection, pes anserine bursitis, neurogenic or vascular claudication, or uncontrolled diabetes mellitus (HbA1C>8%)
* Diagnosis of arthritis due to traumatic injury or meniscal tear in the index knee within 2 years of screening
* Moderate or large knee effusion in the index knee at screening and at test agent administration that requires drainage for diagnostic purposes or symptomatic relief
* Clinically significant, ongoing illness or medical condition that in the opinion of the investigator constitutes a safety risk for participation in the study or that could interfere with achieving the study objectives, conduct or evaluation
* Females who are pregnant or lactating
* Regular use of anticoagulants (daily use of aspirin ≦ 325 mg is acceptable)
* Active alcohol or substance abuse or any other reason that makes it unlikely that the subject will comply with study procedures
* Subjects with a psychiatric illness or condition, which, in the opinion of the investigation, would interfere with the conduct of the study or the interpretation of study results. Subjects with stable anxiety and depression defined as being on stable doses of antidepressant and anxiety drugs for the last 6 months and for which no dose changes are expected during the study can be included.
* Clinically significant medical, surgical, psychiatric, or laboratory abnormality that, in the judgment of the investigator, is likely to adversely affect the subject's risk-benefit or interfere with study compliance or assessment of safety or efficacy.
* Known allergy to local anesthetics or components of the study drug.
* Subjects with autoimmune disease or a known history of having Acquired Immunodeficiency Syndromes (AIDS) or Human Immunodeficiency Virus (HIV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of Signature Cord Prime as defined per CTCAE v. Stopping criteria as defined in 6.11.2.8 | 7 days
  Administered as a single intra-articular injection in subjects with osteoarthritis of knee at 2 dose levels; 75mg and 150mg
Evaluate the safety and tolerability of Signature Cord Prime as defined per CTCAE v. Stopping criteria as defined in 6.11.2.8 | 30 days
  Administered as a single intra-articular injection in subjects with osteoarthritis of knee at 2 dose levels; 75mg and 150mg
Evaluate the safety and tolerability of Signature Cord Prime as defined per CTCAE v. Stopping criteria as defined in 6.11.2.8 | 90 days
  Administered as a single intra-articular injection in subjects with osteoarthritis of knee at 2 dose levels; 75mg and 150mg

SECONDARY OUTCOMES:
Exploratory objective to observe for early data suggestive of efficacy by estimating and comparing changes from baseline | 90 days and six months
  Changes are the differences from the baseline:
  Changes in overall WOMAC Score (WOMAC)
Exploratory objective to observe for early data suggestive of efficacy by estimating and comparing changes from baseline | 90 days and six months
  Changes are the differences from the baseline:
  Changes in overall KOOS Score (KOOS)
Exploratory objective to observe for early data suggestive of efficacy by estimating and comparing changes from baseline | 90 days and six months
  Changes are the differences from the baseline:
  Changes in patient-reported outcomes (PROs) (PROMIS-29)
Exploratory objective to observe for early data suggestive of efficacy by estimating and comparing changes from baseline | 90 days and six months
  Changes are the differences from the baseline:
  Changes in the Pain Visual Analog Scale (100 mm VAS)
Exploratory objective to observe for early data suggestive of efficacy by estimating and comparing changes from baseline | 90 days and six months
  Changes are the differences from the baseline:
  Use of opioid analgesic during study for the affected knee

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Klootwyk, MD, Principal Investigator — Forte Sports Medicine and Orthopedics

IPD SHARING:
Plan to Share IPD: No
Data is proprietary to the manufacturer and will not be shared outside of journal publications.